CLINICAL TRIAL: NCT01952483
Title: Effect of Vitamin D Replacement on Immune Function and Cognition in MS Patients
Status: Completed | Type: Observational
Sponsor: American University of Beirut Medical Center (Other)
Responsible Party: Principal Investigator, Samia Khoury, Professor, American University of Beirut Medical Center
Other Study IDs: IM.SK1.04
Record Dates: First submitted 2013-09-19; First posted 2013-09-30 (Estimated); Last update posted 2018-01-11 (Actual); Status verified 2018-01

CONDITIONS: Multiple Sclerosis (MS)
Keywords: Multiple Sclerosis (MS)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: Samples Without DNA — We will focus on proliferation and cytokine production to myelin basic protein (MBP) and myelin oligodendrocyte glycoprotein (MOG) peptides and on the percentage of Th1 (IFN gamma producing cells) and Th17 (IL-17 producing cells) during in vitro polarization assays
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- vitamin D deficient,: Vitamin D deficiency (serum level <20ng/ml)
- Vitamin D normal: Serum level >35 ng/ml

SUMMARY:
Assessing the immune activation in MS patients deficient in Vitamin D and whether Vitamin D supplementation reverse the immune activation

Evaluating whether Vitamin D deficiency result in lower cognitive performance in MS patients and the effect of Vitamin D supplementation on reversing the cognitive impairment?

DETAILED DESCRIPTION:
We will compare the immune responses in patients with Vitamin D deficiency (serum level <20ng/ml) to those of patients with normal Vitamin D (serum level >35 ng/ml). We will focus on proliferation and cytokine production to myelin basic protein (MBP) and myelin oligodendrocyte glycoprotein (MOG) peptides and on the percentage of Th1 (IFN gamma producing cells) and Th17 (IL-17 producing cells) during in vitro polarization assays. Our hypothesis is that patients with low Vitamin D have increase proliferation to MBP and MOG and increased production of pro-inflammatory cytokines (IFN gamma and IL-17) and that Vitamin D supplementation will decrease this pro-inflammatory profile.

We will measure cognitive performance in patients with Vitamin D deficiency (serum level <20ng/ml) compared to those of patients with normal Vitamin D (serum level >35 ng/ml) after adjusting for educational levels and disease duration. We hypothesize that low Vitamin D has a negative effect on cognitive performance and that Vitamin D supplementation will improve cognitive function.

ELIGIBILITY:
Inclusion Criteria:

1. Definite diagnosis of Multiple Sclerosis following the revised McDonald MS diagnostic criteria
2. Male and Female Aged 18 and above
3. On interferon-β treatment (Rebif®, Avonex®, or Betaseron®)
4. No signs of active inflammation or attack or new lesions on MRI

Exclusion Criteria:

1. Treatment with immune modulating/ suppressive drugs other than IFN-b within 6 weeks prior to enrolment
2. Pregnancy
3. Hypercalcemia
4. eglomerular filtration rate<60
5. History of primary hyperparathyroidism, hypercalcemia, renal dysfunction, cardiac disease, malignancy, or granulomatous disease
6. The occurrence of an exacerbation (defined as an episode of neurologic dysfunction lasting at least 24 hours) within 4 weeks of enrollment
7. History of dementia or related disorders
8. History of traumatic brain injury
9. Diagnosis of epilepsy or history of seizure
10. Diagnosis of psychiatric disease, substance abuse/dependence, alcohol abuse/dependence
11. Currently, on any of the following medications Lithium, or Thiazide diuretics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Group 1: low vitamin D (less than 25 ng/ml) Group 2: normal vitamin D level (greater than 35 ng/ ml)
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2012-08; Primary Completion 2017-05-01 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Is there evidence of immune activation in MS patients deficient in Vitamin D and does Vitamin D supplementation reverse the immune activation? | 3months
  We will compare the immune responses in patients with Vitamin D deficiency (serum level <20ng/ml) to those of patients with normal Vitamin D (serum level >35 µg/ml). We will focus on proliferation and cytokine production to myelin basic protein (MBP) and myelin oligodendrocyte glycoprotein (MOG) peptides and on the percentage of Th1 (IFN gamma producing cells) and Th17 (IL-17 producing cells) during in vitro polarization assays. Our hypothesis is that patients with low Vitamin D have increase proliferation to MBP and MOG and increased production of pro-inflammatory cytokines (IFN gamma and IL-17) and that Vitamin D supplementation will decrease this pro-inflammatory profile.

SECONDARY OUTCOMES:
Does Vitamin D deficiency result in lower cognitive performance in MS patients and does Vitamin D supplementation reverse the cognitive impairment? | 3 months
  We will measure cognitive performance in patients with Vitamin D deficiency (serum level <20ng/ml) compared to those of patients with normal Vitamin D (serum level >35 ng/ml) after adjusting for educational levels and disease duration. We hypothesize that low Vitamin D has a negative effect on cognitive performance and that Vitamin D supplementation will improve cognitive function.

CONTACTS AND LOCATIONS:
Overall Officials: Samia J Khoury, professor, Principal Investigator — AUBMC
Locations (1):
- AUBMC Multiple Sclerosis Center, Beirut, Riad El Solh, Lebanon

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Khoo AL, Joosten I, Michels M, Woestenenk R, Preijers F, He XH, Netea MG, van der Ven AJ, Koenen HJ. 1,25-Dihydroxyvitamin D3 inhibits proliferation but not the suppressive function of regulatory T cells in the absence of antigen-presenting cells. Immunology. 2011 Dec;134(4):459-68. doi: 10.1111/j.1365-2567.2011.03507.x. PMID 22044285
- [Background] Zivadinov R, Sepcic J, Nasuelli D, De Masi R, Bragadin LM, Tommasi MA, Zambito-Marsala S, Moretti R, Bratina A, Ukmar M, Pozzi-Mucelli RS, Grop A, Cazzato G, Zorzon M. A longitudinal study of brain atrophy and cognitive disturbances in the early phase of relapsing-remitting multiple sclerosis. J Neurol Neurosurg Psychiatry. 2001 Jun;70(6):773-80. doi: 10.1136/jnnp.70.6.773. PMID 11385012
- [Background] Adorini L, Penna G, Giarratana N, Roncari A, Amuchastegui S, Daniel KC, Uskokovic M. Dendritic cells as key targets for immunomodulation by Vitamin D receptor ligands. J Steroid Biochem Mol Biol. 2004 May;89-90(1-5):437-41. doi: 10.1016/j.jsbmb.2004.03.013. PMID 15225816
- [Background] Przybelski RJ, Binkley NC. Is vitamin D important for preserving cognition? A positive correlation of serum 25-hydroxyvitamin D concentration with cognitive function. Arch Biochem Biophys. 2007 Apr 15;460(2):202-5. doi: 10.1016/j.abb.2006.12.018. Epub 2007 Jan 8. PMID 17258168
- [Background] Barake M, Daher RT, Salti I, Cortas NK, Al-Shaar L, Habib RH, Fuleihan Gel-H. 25-hydroxyvitamin D assay variations and impact on clinical decision making. J Clin Endocrinol Metab. 2012 Mar;97(3):835-43. doi: 10.1210/jc.2011-2584. Epub 2012 Jan 11. PMID 22238386